CLINICAL TRIAL: NCT03215862
Title: The Effect of the Use of Lactated Ringer's Solution During ERCP on Rate of Post-endoscopic Retrograde Cholangiopancreatography (ERCP) Pancreatitis
Brief Title: Lactated Ringer's Solution to Prevent Post-ERCP Pancreatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00029546
Record Dates: First submitted 2017-07-10; First posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: Post-ERCP Acute Pancreatitis; Normal Saline; Lactated Ringer's
MeSH Terms: interventions — Ringer's Lactate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Drug: Normal Saline 0.9% Infusion Solution Bag
- Experimental (Experimental)
  Interventions: Drug: Lactated Ringer

INTERVENTIONS:
Drug: Lactated Ringer — This is a Lactated Ringer's solution infusion before, during, and after the ERCP procedure.
  Arms: Experimental
Drug: Normal Saline 0.9% Infusion Solution Bag — This is a Normal Saline solution infusion before, during, and after the ERCP procedure.
  Arms: Control

SUMMARY:
This is a randomized, double-blinded, controlled trial. This study is a head to head comparison of normal saline (NS) infusion versus Lactated Ringer's (LR) infusion in patients, with the primary outcome of post-ERCP pancreatitis occurrence. Patients will be randomized to either the NS infusion group or the LR infusion group. IVF will be started pre-procedurally and will be continued throughout the procedure. A IVF bolus will be given at the end of the procedure and then continued as a continuous infusion. Our null hypothesis is that there will be no significant difference in the rate of occurrence of post-ERCP pancreatitis between the infusion of LR and NS solutions. Our alternative hypothesis is that patients receiving LR solution infusion will experience a decreased rate of post-ERCP pancreatitis compared to patients receiving NS solution infusion.

ELIGIBILITY:
Inclusion Criteria:

i. Possession of one of the following criteria which places the patient at high risk for post-ERCP pancreatitis and/or if patient is to undergo a planned endoscopic intervention deemed at high risk:

1. Suspicion of Oddi dysfunction
2. Personal history of post-ERCP pancreatitis
3. More than 8 cannulation attempts
4. Precut sphincterotomy
5. Endoscopic papillary balloon dilation of an intact sphincter
6. Endoscopic pancreatic duct sphincterotomy
7. Ampullectomy
8. Total bilirubin < 1.0

ii. Or possession of two or more of the following minor criteria:

1. Female sex
2. Age under 50 years
3. Personal history of recurrent acute pancreatitis
4. Pancreatic duct injection leading to "acinarization" or over 3 pancreatic duct injections
5. Pancreatic duct cytology acquisition

Exclusion Criteria:

1. Patients aged less than 18
2. Inability to provide informed consent
3. Pregnancy
4. Active acute pancreatitis
5. Any contraindication to aggressive IVF hydration: evidence of clinical volume overload (peripheral or pulmonary edema), respiratory compromise (oxygen saturation < 90% on room air), chronic kidney disease (creatinine clearance < 40 mL/min), systolic congestive heart failure (ejection fraction < 45%), cirrhosis, and severe electrolyte disturbance with sodium <130 mEq/L or >150 mEq/L
6. If patient does not undergo a planned high-risk intervention
7. If patient does not possess complete criteria which places them at high risk for post-ERCP pancreatitis
8. Patients with cholangitis
9. Patients with chronic and/or active pancreatitis
10. Patients with a true NSAID allergy
11. Patients greater than or equal to 75 years old

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Post-ercp pancreatitis | 24 hours
  The occurrence of pancreatitis as a complication of ERCP procedure, assessed 24 hours after the procedure is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Pushpak Taunk, MD, Principal Investigator — University of South Florida

IPD SHARING:
Plan to Share IPD: No